CLINICAL TRIAL: NCT02108938
Title: Characterizing Brain-Gut Interaction in Patients With Crohn's Disease Using Advanced Neuroimaging Tools
Brief Title: Brain-Gut Interactions in Crohn's Disease
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0131
Record Dates: First submitted 2014-03-24; First posted 2014-04-09 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Subject's with Crohn's disease at least 18 years of age
- Control: Findings from this study will be compared to "controls." These controls will come from the well documented CNS changes which have been found in patients with IBS and chronic pancreatitis (HS-IRB# 2013-1561 and HS-IRB 2009-0171).

SUMMARY:
The primary aims for this research are to 1) characterize brain changes in patients with CD compared to age and gender-matched controls and 2) relate these brain changes to measures of disease activity and pain severity.

DETAILED DESCRIPTION:
Brain-gut interactions have been studied in chronic pain conditions of the gastrointestinal (GI) tract such as irritable bowel syndrome (IBS) and chronic pancreatitis. These studies suggest that alterations in the brain-gut axis may relate to disease severity and pain perception. Inflammatory bowel disease (IBD) is a chronic inflammatory disorder characterized by periods of disease activity and periods of disease quiescence. Crohn's disease (CD) is one of the two major subtypes of IBD. Patients with CD typically experience abdominal pain when the disease is active; however, many also report experiencing pain in the absence of objective evidence of inflammation. Alterations in brain-gut interactions may explain the perception of pain in these patients. Currently, there is a paucity of data regarding brain changes in patients with IBD and CD, specifically. We are proposing a pilot study to characterize brain-gut interactions of disease activity and pain modulation mechanisms in patients with IBD using advanced neuroimaging tools.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* A diagnosis of Crohn's disease by endoscopy or radiographic imaging
* Must have Crohn's disease in symptomatic remission as defined by a Harvey-Bradshaw score of 3
* No contraindications to MRI per UWHC screening form
* Able to provide informed consent

Exclusion Criteria:

* Women that are pregnant
* Contraindications to MRI per UWHC screening form
* Other chronic pain disorders (e.g. fibromyalgia, rheumatoid arthritis, irritable bowel disorder) unrelated to their diagnosis of IBD.
* Scheduled medications for the treatment of pain (e.g. acetaminophen, non-steroidal anti-inflammatory drugs, narcotics) will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older diagnosed with CD, as determined by endoscopy or radiographic imaging, will be targeted for enrollment. Patients with CD in symptomatic remission as defined by a Harvey-Bradshaw score of 3, will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2015-05-18 (Actual); Study Completion 2015-05-18 (Actual)

PRIMARY OUTCOMES:
1) characterize brain changes in patients with CD compared to age and gender-matched controls | 1 year
  Because of the relatively large number of predictor variables in relation to the potential number of subjects, these analyses will be considered exploratory and aimed at generating hypotheses. Future studies with a larger number of subjects can be focused on hypothesis-driven questions and in developing diagnostic brain-based biomarkers and determining whether novel treatments aimed at the brain-gut axis may alter disease activity and pain perception in this patient population.

SECONDARY OUTCOMES:
2) relate these brain changes to measures of disease activity and pain severity. | 1 year
  Because of the relatively large number of predictor variables in relation to the potential number of subjects, these analyses will be considered exploratory and aimed at generating hypotheses. Future studies with a larger number of subjects can be focused on hypothesis-driven questions and in developing diagnostic brain-based biomarkers and determining whether novel treatments aimed at the brain-gut axis may alter disease activity and pain perception in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Sumona Saha, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital & Clinics, Madison, Wisconsin, United States